CLINICAL TRIAL: NCT01752465
Title: Is Health Coaching a Useful Clinical Tool to Facilitate Healthy Lifestyle Change and Improve Metabolic Health in People With Psychotic Illness?
Brief Title: Is Health Coaching Effective for Improving Metabolic Health in People With Psychosis Disorders?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H12-01896; F12-01992 (Other: UBC Office of Research Services)
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Psychotic Disorders; Metabolic Syndrome x
Keywords: Health behaviour; Antipsychotic agents; Adverse effects; Goals; Life style
MeSH Terms: conditions — Psychotic Disorders; Metabolic Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): Patients in the standard care group will receive standard clinical care from their attending psychiatrist, including pharmacotherapy and education. Study assessments will be done at baseline, and once a month thereafter at Months 1, 2, 3, and 6.
  Interventions: Behavioral: Health Coaching; Behavioral: Standard care
- Health Coaching (Experimental): Patients in the Health Coaching group will receive both Health Coaching, and standard care. In addition to routine clinical appointments, patients receiving Health Coaching will attend Health Coaching sessions twice a month during Months 1, 2, and 3, and once a month during Months 4, 5, and 6. Study assessments will be conducted at baseline, and once a month thereafter during Health Coaching sessions at Months 1, 2, 3, and 6.
  Interventions: Behavioral: Health Coaching

INTERVENTIONS:
Behavioral: Health Coaching — Health Coaching sessions are 2 hours long. Participants individually receive a physical assessment, and recent blood work and medications are reviewed. When everyone has been assessed, the group reconvenes to watch a video about the importance of making healthy lifestyle choices, participates in a 10 min. fitness activity, and receives training on making SMART goals (SMART stands for specific, measurable, achievable, realistic, and timely). Each participant individually creates a SMART goal for him/herself, and this goal is reviewed as a group. Each participant rates the importance of this goal, and rates their level of confidence in succeeding. Progress is tracked in subsequent sessions, and metabolic health is continually monitored through routine blood work.
  Other Names: Integrative Health Coaching; EPI Metabolic Group
Behavioral: Standard care — Standard clinical care will continue for all participants in the study, regardless of the study arm. This includes routine clinical visits to the attending psychiatrist, and receiving pharmacotherapy, standard patient education, and psychosocial training.
  Arms: Standard Care

SUMMARY:
Antipsychotic medications frequently cause metabolic side-effects, such as abdominal obesity, high blood pressure, cholesterol abnormalities, and blood sugar dysregulation, all of which can lead to what is known as the Metabolic Syndrome and serious long-term cardiovascular health problems. Therefore, it is important that metabolic issues be addressed as part of a holistic approach to the mental health treatment of these patients.

As with the general population, improving metabolic health involves lifestyle changes - i.e., addressing daily habits regarding eating, physical exercise, stress and sleep management, and lifestyle habits such as smoking. However, there is growing recognition in the medical field that education is not enough for people to create meaningful and sustained lifestyle change. The emerging field of Integrative Health Coaching addresses this issue and provides a clinical framework for helping people successfully develop and achieve personalized lifestyle goals. The investigators have therefore decided to investigate whether health coaching techniques may have benefit in addressing metabolic health issues in people with psychosis disorders. The intent is to complement usual psychiatric and medical care, and also promote patient engagement in managing one's overall health.

This study will investigate whether Integrative Health Coaching is a useful clinical tool to facilitate healthy lifestyle behaviour and thereby improve metabolic health in people with psychosis disorders.

DETAILED DESCRIPTION:
Antipsychotic drugs are widely used to treat not only psychosis but an increasing number of other psychiatric indications. The prevalence of antipsychotic drug use in British Columbia is increasing at a high rate, especially in youth. Second generation ("atypical") antipsychotic drugs, while bereft of the neurological side-effects of their predecessors, commonly cause metabolic syndrome. This includes hyperglycemia, hyperlipidemia, insulin resistance, weight gain and hypertension - a cluster of side-effects that puts patients at strongly increased risk of cardiometabolic disorders such as Type 2 diabetes and cardiovascular disease. Drug therapies to reduce metabolic dysregulation have provided limited benefits. It is recognized that lifestyle changes that address daily habits regarding eating, physical exercise, stress and sleep management, and lifestyle habits such as smoking, represent a complementary approach to additional drug therapy. The emerging field of Integrative Health Coaching addresses this issue and provides a clinical framework for helping people successfully develop and achieve personalized lifestyle goals. This study will investigate whether Health Coaching is a useful clinical tool to facilitate healthy lifestyle behavior and thereby improve metabolic health in people with psychotic illness.

HYPOTHESIS: In a first-episode psychosis population that have recently begun treatment with atypical antipsychotic drugs, the inclusion of an Integrative Health Coaching goal-setting model will significantly improve patients' attitudes towards, and increase the frequency of behaviours related to healthy living, as indicated by the Short-Form 36, the Three-Factor Eating Questionnaire, and the Health Value Scale.

RESEARCH PLAN: The investigators will conduct a non-blinded clinical trial of the efficacy of Integrative Health Coaching techniques in 40 subjects who are being treated at the Vancouver/Richmond Early Psychosis Intervention program, which provides specialty care to patients with suspected or newly diagnosed psychotic disorders. All subjects will be randomly assigned to one of two treatment groups (n = 20 subjects per group). In the first group, subjects will receive treatment for psychosis based on the current standard of care, which includes psychosocial training, education and pharmacological treatment. The second group of subjects will receive not only the standard of care treatment for psychosis, but additional Health Coaching to improve physical health. Subjects in both treatment groups will be given questionnaires to assess health attitudes and behaviours, and will receive routine blood work to monitor metabolic dysregulation, at baseline and months 1, 2, 3 and 6 from when they enter the study. Data will be collected and analyzed for differences between the two groups at the end of the study. Results will be analyzed based on intent-to-treat analysis, and comparison of metabolic and other health indices compared between the two groups using t-test and chi-square analyses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a primary working diagnosis of schizophrenia/schizoaffective disorder, or bipolar disorder, or psychosis not otherwise specified (PNOS)
* Subjects must be prescribed an atypical (or 'second-generation') antipsychotic drug

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Scores on the Short-Form 36 | Baseline, month 1, month 2, month 3, and month 6
  Scores on the Short-Form 36 (a standardized, validated questionnaire measuring general health) will be compared between patients in the Health Coaching group versus patients receiving only standard care.
Scores on The Three Factor Eating Questionnaire (TFEQ) | Baseline, month 1, month 2, month 3, and month 6
  Scores on the Three Factor Eating Questionnaire (a questionnaire measuring cognitive restraint of eating, disinhibition, and hunger) will be compared between patients in the Health Coaching group, versus patients receiving only standard care.
Scores on The Health Value Scale | Baseline, month 1, month 2, month 3, and month 6
  Scores on the Health Value Scale (a questionnaire measuring value placed on health) will be compared between patients in the Health Coaching group, versus patients receiving standard care only.

SECONDARY OUTCOMES:
Waist circumference | Baseline, month 1, month 2, month 3, and month 6
  Change in waist circumference over 6 months, and comparison of the change in waist circumference between patients in the Health Coaching group, versus patients receiving standard care only.
Blood Pressure | Baseline, month 1, month 2, month 3, and month 6
  Change in systolic and diastolic blood pressure over 6 months, and comparison of the change in systolic and diastolic blood pressure between patients receiving Health Coaching, and patients receiving standard care only.
Heart Rate | Baseline, month 1, month 2, month 3, and month 6
  Change in heart rate over 6 months, and comparison of the change in heart rate between patients receiving Health Coaching, versus patients receiving standard care only.
Fasting plasma glucose | Baseline, month 1, month 2, month 3, and month 6
  Change in fasting plasma glucose over 6 months, and comparison of the change in fasting plasma glucose between patients in the Health Coaching group, versus patients receiving standard care only.
Fasting total cholesterol | Baseline, month 1, month 2, month 3, and month 6
  Change in fasting total cholesterol over 6 months, and comparison of the change in fasting total cholesterol between patients in the Health Coaching group, versus patients receiving standard care only.
Fasting cholesterol subfractions | Baseline, month 1, month 2, month 3, and month 6
  Change in fasting cholesterol subfractions (LDL-C, HDL-C) over 6 months, and comparison of the change in fasting cholesterol subfractions between patients receiving Health Coaching, versus patients receiving standard care only.
Fasting triglycerides | Baseline, month 1, month 2, month 3, and month 6
  Change in fasting triglycerides over 6 months, and comparison of the change in fasting triglycerides between patients receiving Health Coaching, versus patients receiving standard care only.
Fasting insulin | Baseline, month 1, month 2, month 3, and month 6
  Change in fasting insulin over 6 months, and comparison of the change in fasting insulin between patients receiving Health Coaching, versus patients receiving standard care only.

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair M Barr, Ph.D., Principal Investigator — The University of British Columbia
Locations (1):
- Vancouver/Richmond Early Psychosis Intervention Clinic, Vancouver, British Columbia, Canada